CLINICAL TRIAL: NCT04369651
Title: Socio-economic Determinants for Acceptance and Choice of Biological Treatment by Patients With Spondyloarthropathy in Nepal
Brief Title: Socio-economic Determinants for Acceptance and Choice of Biological Treatment
Status: Completed | Type: Observational
Sponsor: National Center for Rheumatic Diseases, Nepal (Other)
Responsible Party: Principal Investigator, Shweta Nakarmi, Study coordinator, National Center for Rheumatic Diseases, Nepal
Other Study IDs: 210/2017
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Spondyloarthritis
Keywords: socio-economic determinants; biologic; Nepal; low income country; spondyloarthroathy
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This was a cross-sectional study conducted at National center for rheumatic diseases, Nepal on SpA patient refractory to initial treatment with conventional anti rheumatic drugs. Patients taking TNFi (tumor necrosis factor inhibitor- adalimumab or etanercept) or tofacitinib were included. Baseline demographic, socio-economic, clinical data were recorded.

DETAILED DESCRIPTION:
This was a cross-sectional observational study conducted in the rheumatology clinic of National Center for Rheumatic Diseases, Kathmandu, Nepal. Patients with spondyloarthropathy (SpA) and enrolled in the cohort database from June 2015 to December 2019 were selected. Those taking any oral or injectable forms of biological treatment were included in the study. Patients less than 18 years of age, who did not consent for participation or additional information, who were deferred from biological treatment due to comorbid conditions like concurrent infections or heart failure were excluded. An informed consent was obtained from selected patients and any additional information required was taken via e-mail or telephone enquiry.

Diagnostic & measurement tools Diagnosis of SpA was made by rheumatologists on the basis of the modified New York Criteria for Ankylosing Spondylitis and the ASAS criteria (Assessment of SpondyloArthritis International Society) for axial and peripheral SpA. Diagnosis of nr-axial SpA was made by MRI evidence of sacroilitis in a patient with normal radiograph with or without HLA B27. Disease activity was assessed using composite Ankylosing Spondylitis Disease Activity Score (ASDAS) and the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI).

Socioeconomic status Socioeconomic factors studied were educational level and the primary occupation. Patient self-reported highest educational level was recorded and was categorized into illiterate, primary, secondary, higher secondary, above secondary level education. Occupation and social class were recorded based on self-report primary source of income. It was categorized into homemakers, students, service holders, business, teachers, farmers and others (field workers, labor workers). A dedicated research officer also took data on other demographic parameters and geographical location of residence. Geographical location was categorized into urban-rural and hilly-plain terrain.

Indications for offering biological treatment Indications for biological or small molecule treatment included: a. Failure of at least 2 courses of NSAIDS, b. Failure of at least 3months of conventional synthetic DMARDs (csDMARDs). For patients with PsA, the csDMARDs included methotrexate and/or leflunomide; for AS, nr-axial SpA and IBD-associated arthritis, it included sulfasalazine and/or methotrexate. Failure of treatment was defined as: a. Persistent ASDAS of ≥2.1, b. Improvement of ASDAS by less than -1.1, c. Persistent BASDAI of ≥4. All patients fulfilling these indications were offered biological treatment. Patients with no contraindication for TNFi were offered either injectable biologicals (adalimumab or etanercept: only TNFi available in Nepal) or tofacitinib (only small molecule available in Nepal) and explained about the preparatory investigations, dosage of TNFi, storage, cost, monitoring and side-effects.

Data collection and analysis Complete data on baseline demographic parameters (age, gender, address, education, occupation) and ASDAS and BASDAI scores at initiation of treatment with biological or small molecule were recorded in a hardcopy data-sheet and later entered to a predesigned excel-sheet by a trained research officer.

Statistical analysis was performed using SPSS version 21 (IBM Corp, USA). Simple descriptive statistics were used to analyze various socioeconomic and demographic parameters. Chi-squared test was used to analyze difference in these parameters between patients who chose injectable and those who chose tofacitinib. Linear regression analysis was performed to identify variables associated with use of any biological agent. All variables with p-value of <0.05 were analyzed in multiple regression model to evaluate the independent association. Difference in mean values between two treatment groups were assessed by independent t-test.

ELIGIBILITY:
Inclusion Criteria:

* patients with spondyloarthropathy
* on any oral or injectable forms of biological treatment

Exclusion Criteria:

* less than 18years of age
* who did not consent for participation
* deferred from biological treatment due to comorbid conditions like concurrent infections or heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SpA and enrolled in the cohort database from June 2015 to December 2019 were selected.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
socio economic determinants | four years
  socio economic determinants for acceptance of biologic therapy

IPD SHARING:
Plan to Share IPD: Undecided